CLINICAL TRIAL: NCT04318028
Title: A Pilot Study of 7 Tesla MRI Neuroimaging Biomarkers of Prostate Cancer-Related Cognitive Impairment
Brief Title: An Investigational Scan (7 Tesla MRI) in Diagnosing Cognitive Impairment in Patients With Non-Metastatic Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4P-19-4; NCI-2019-05018 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4P-19-4 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Non-Metastatic Prostate Carcinoma; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (7 Tesla MRI) (Experimental): Patients undergo 7 Tesla MRI over 30-90 minutes at baseline and 6-9 months.
  Interventions: Procedure: 7 Tesla Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: 7 Tesla Magnetic Resonance Imaging — Undergo 7 Tesla MRI
  Other Names: 7 Tesla MRI; 7T MRI

SUMMARY:
This trial studies 7 Tesla magnetic resonance imaging (MRI) in diagnosing cognitive impairment in patients with prostate cancer that has not spread to other places in the body (non-metastatic) and who have or have not received androgen deprivation therapy (ADT). The MRI machine uses a strong magnet and radio wave to make images of the inside of the body. A stronger magnetic field allows greater signals and more detailed visualization of the structure and function of human body. Giving 7 Tesla MRI may help doctors learn if patients that receive ADT show more signs of cognitive dysfunction or brain fog compared to patients to patients that do not receive ADT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Observe longitudinal changes in structural connectivity using T1-weighted and diffusion tensor MRI in men with non-metastatic prostate cancer on current ADT versus those who were not.

II. Observe longitudinal changes in brain functional connectivity using resting-state functional (rsf) MRI.

III. Observe longitudinal changes in brain metabolic profiles evaluated by MR spectroscopy (MRS).

IV. Exploratory assessment of correlation between testosterone and prostate specific antigen (PSA) levels with MRI measures and cognitive measures.

SECONDARY OBJECTIVES:

I. To assess the feasibility and acceptability of this approach using sequential 7T MRI in prostate cancer patients either receiving ADT or not.

OUTLINE:

Patients undergo 7 Tesla MRI over 30-90 minutes at baseline and at 6-9 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent
* Group 1 (G1): Non-metastatic biopsy-proven prostate cancer patients on current ADT and
* Group 2 (G2): Demographically (age, cancer stage) matched non-metastatic biopsy proven prostate cancer patients without a history of ADT
* Ability to undergo imaging procedure without any form of sedation
* Ability to complete brief cognitive testing on iPad

Exclusion Criteria:

* History of dementia or other neuropsychiatric disease
* History of other cancer medical therapies other than ADT, narcotics or psychiatric medications
* Standard contraindications for MRI:

  * Prior work as a machinist or metal worker, or history of metal being removed from the eyes,
  * Cardiac pacemaker or internal pacing wires,
  * Non-MRI compatible vena cava filter, vascular aneurysm clip, heart valve, spinal or ventricular shunt, optic implant, neuro-stimulator unit, ocular implant, or intrauterine device, or
  * Claustrophobia, or uncontrollable motion disorder
* Currently active second malignancy
* Any significant cardiovascular conditions (New York Heart Association [NYHA]) class III or IV congestive heart failure, myocardial infarction within 6 months, unstable angina, pacemaker); or
* Renal disease with calculated creatinine clearance of < 45 ml/min

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Brain structural connectivity | Up to 1 year
  Will be measured using T1-weighted and diffusion tensor magnetic resonance imaging (MRI).
Brain functional connectivity | Up to 1 year
  Will be measured using resting-state functional MRI.
Brain metabolic profiles | Up to 1 year
  Will be evaluated by MR spectroscopy.

OTHER OUTCOMES:
Assessment of testosterone and prostate specific antigen (PSA) levels | Up to 1 year
  For the correlation of between testosterone and PSA levels with MRI measures and cognitive measures, the study will use scatter plots to explore the pattern of correlation. Spearmen's correlation will be used to test the correlation. Both groups will be combined for the correlation analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Shiroishi, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States